CLINICAL TRIAL: NCT00331435
Title: Clinical Research of Photodynamic Therapy for Exudative Age-related Macular Degeneration Accompanied With Polypoidal Choroidal Vasculopathy
Brief Title: PDT Study for Exudative AMD With PCV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ophthalmic PDT Study Group (Other)
Responsible Party: Tomohiro Iida, Ophthalmic PDT study group
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCV-PDT-1
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD; PCV; PDT
MeSH Terms: conditions — Macular Degeneration | interventions — Verteporfin; Photochemotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): FA-guided PDT
  Interventions: Procedure: Ocular photodynamic therapy with verteporfin
- 2 (Experimental): ICG-guided PDT
  Interventions: Procedure: Ocular photodynamic therapy with verteporfin

INTERVENTIONS:
Procedure: Ocular photodynamic therapy with verteporfin — Ocular photodynamic therapy with 6 mg per meter squar of body sarface of verteporfin with PDT lazer application for 83 seconds
  Other Names: photodynamic therapy

SUMMARY:
The purpose of this study is to evaluate and conduct an exploratory comparison of the efficacy and safety of indocyanine green angiography (ICGA) guided photodynamic therapy (PDT) and fluorescein angiography (FA) guided PDT for exudative age-related macular degeneration (AMD) accompanied with polypoidal choroidal vasculopathy (PCV).

DETAILED DESCRIPTION:
PDT with verteporfin has been proven beneficial for patients with AMD. The laser spot size is decided based on FA finding (FA guided PDT). ICGA is needed to detect PCV lesions, such as polypoidal lesions or abnormal network vessels. In clinical practice, PDT based on ICGA (ICGA guided PDT) has and is being conducted for the treatment of AMD with PCV. However, there are no reports on the outcomes of prospective research of PDT for PCV in Japanese patients. Furthermore, there are no reports comparing FA guided PDT and ICGA guided PDT.

We propose to conduct this clinical research in order to investigate the efficacy and safety of PDT for PCV in Japanese patients, and to compare results of FA guided PDT and ICGA guided PDT.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients aged 50 years old or older
* Exudative AMD with subfoveal PCV
* Eyes with PCV meets the definite criteria of PCV issued from Japanese study group of Polypoidal Choroidal Vasculopathy
* PCV lesion with subfoveal hemorrhage or exudation
* Lesion size (GLD) of less than 12 MPS Disc area measured by FA and IA.
* Decimal BCVA of 0.1-0.5 at baseline period.

Exclusion Criteria:

* Patients who have RPE tear, vitelliform retinal dystrophy, and central Serous Chorioretinopathy.
* Patients who have other ocular disease with irreversible VA
* Study eyes unable to be taken fundus photos of CNV
* Study eyes received surgery operation within 2 months of the participation to this study or ND:YAG operation within one month
* Pathological myopia
* PCV with cleary identified subsensory retinal CNV (on the RPE) at the baseline examination
* Study eyes which have received any treatments for CNV, such as PDT, transpupillary thermotherapy, laser photocoagulation, and so on.
* Patients who have any physical problem for using angiography or PDT (such as systemic debility, significant diabetes mellitus, significant heart disease, and so on)
* Medical history of porphyria, porphyrin sensitivity, or hypersensitivity to sunlight or bright light.
* Patients with medical history of hypersensitivity to ingredients of Visudyne
* Patients with medical history of hypersensitivity to ingredients of fluorescein or indocyanine green injection
* Patients with hypersensitivity to iodine
* Patients judged inappropriate for this study by the investigator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Proportion of study eyes which best corrected visual acuity (BCVA) improves 2 lines or more or maintains (+/-1 line changes) at 12 months after first treatment, as compared with the visual acuity at baseline period. | 12 months

SECONDARY OUTCOMES:
Proportion of number of study eyes which BCVA improves 3 lines or more or maintains (+/-1 line), as compared with baseline examination. | 12 month
Factor affecting to change in visual acuity. | 12month
Proportion of eyes with decimal BCVA of 0.5 or more. | 12 month
Change of findings of polypoidal lesions. | 0-12 month
Change of findings of abnormal network vessels. | 0-12 month
Change in greatest linear dimension (GLD) based on FA. | 0-12 month
PCV lesion size based on ICGA. | 0-12 month
Choroidal neovascularization (CNV) closure based on FA. | 0-12 month
Change in subretinal fluid at the fovea and central retinal thickness based on optical coherence tomography (OCT). | 0-12month
Mean number of PDT treatments required during the study period. | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Tomohiro Iida, MD, Principal Investigator — Ophthalmic PDT Study Group
Locations (17):
- Japan (17):
  - Nagoya City University Hospital, Aichi
  - Nagoya University, Aichi
  - Kyushu University, Fukuoka
  - Fukushima Medical University School of Medicine, Fukushima
  - Gunma University, Gunma
  - Kagawa University, Kagawa
  - Kyoto University, Kyoto
  - Osaka University, Osaka
  - Kansai Medical University Takii Hospital, Osaka
  - Kansai Medical University Hirakata Hospital, Osaka
  - Sapporo City general hospital, Sapporo
  - Shiga University of Medical Science, Shiga
  - Surugadai Nihon University Hospital, Tokyo
  - Kyorin University, Tokyo
  - Toho University, Tokyo
  - Tokyo University Ohashi Medical Center, Tokyo
  - Yamanashi University, Yamanashi